CLINICAL TRIAL: NCT03567473
Title: A Randomized Controlled Trial Comparing Epinephrine and Dexamethasone to Placebo in the Treatment of Infants With Bronchiolitis
Brief Title: Bronchiolitis in Infants Placebo Versus Epinephrine and Dexamethasone Study
Acronym: BIPED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital Research Institute of Manitoba (Other); Research Manitoba (Other); Women and Children's Health Research Institute, University of Alberta (Unknown); Alberta Children's Hospital Research Institute (Other); The Hospital for Sick Children (Other); Department of Pediatrics, Western University (Unknown); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Amy Plint, MD, MSc, FRCPC, Research Chair in Pediatric Emergency Medicine, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO 1423
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel (including study nurses, coordinators, investigators, data management staff, and statistical team), health care staff providing patient care, and patients/families will be blinded to the study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Intervention Arm (Experimental): Oral dexamethasone and nebulized epinephrine OR Oral dexamethasone and inhaled epinephrine given by MDI
  Interventions: Drug: Oral dexamethasone; Drug: Nebulized Epinephrine; Drug: MDI Epinephrine
- Control Arm (Placebo Comparator): Oral placebo (OraBlendTM in Canada and a compounded oral placebo solution at New Zealand/Australia sites) and nebulized saline.
  OR Oral placebo (OraBlendTM in Canada and a compounded oral placebo solution at New Zealand/Australia sites) and inhaled placebo given by MDI.
  Interventions: Drug: Oral placebo; Drug: Nebulized normal saline; Drug: MDI placebo

INTERVENTIONS:
Drug: Oral dexamethasone — Two doses of oral dexamethasone, 0.6 mg/kg (maximum single dose 10 mg). One at the time of emergency department enrolment immediately prior to first nebulized treatment and one at approximately 24 hour later
  Other Names: Dexamethasone
  Arms: Active Intervention Arm
Drug: Nebulized Epinephrine — Two nebulized treatments of 3 mL 1:1000 epinephrine 30 minutes apart (+/- 15 minutes) at the time of emergency department enrolment
  Other Names: Nebulized Adrenaline
  Arms: Active Intervention Arm
Drug: Oral placebo — Two doses of oral placebo, 0.6 mL/kg (maximum single dose 10 mL). One at the time of emergency department enrolment immediately prior to nebulized treatment and one at approximately 24 hour later . Oral placebo at Canadian sites is composed of OraBlendTM and in New Zealand and Australian sites will be a compounded solution.
  Other Names: Placebo
  Arms: Control Arm
Drug: Nebulized normal saline — Two nebulized treatments of 3 mL of normal saline 30 minutes apart (+/- 15 minutes) at the time of emergency department enrolment
  Other Names: Saline
  Arms: Control Arm
Drug: MDI Epinephrine — Two doses of Epinephrine given by MDI plus spacer at 625 mcg (5 actuations of 125mcg) 30 minutes apart (+/- 15 minutes) at the time of emergency department enrolment.
  Other Names: MDI Adrenaline
  Arms: Active Intervention Arm
Drug: MDI placebo — Two doses of inhaled placebo given by MDI plus spacer, 30 minutes apart (+/- 15 minutes) at the time of emergency department enrolment.
  Other Names: Placebo
  Arms: Control Arm

SUMMARY:
We hypothesize that infants with bronchiolitis treated with inhaled epinephrine in the Emergency Department (ED) and a 2-day course of oral dexamethasone will have fewer hospitalizations over 7 days compared to infants treated with placebo. To examine this hypothesis, we will conduct a phase III, multicentre, randomized, double-blind trial. Infants presenting to one of twelve study EDs will be enrolled to one of two study groups: (1) inhaled epinephrine and oral dexamethasone or (2) inhaled placebo and oral placebo. Our primary outcome will be admission for bronchiolitis by day 7 following the enrolment. As a planned secondary analysis, a between-group comparison of the primary outcome will be performed in those patients presenting with a first episode of bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to the ED with an episode of bronchiolitis. Bronchiolitis will be defined as an episode of wheezing or crackles in a child < 12 month of age associated with signs of an upper respiratory tract infection (e.g. cough, coryza, nasal congestion) during the period deemed to be peak season for RSV bronchiolitis (approximately December to April in Northern Hemisphere and June to October in Southern Hemisphere). We have chosen not to define bronchiolitis as the first episode of wheezing or crackles to better reflect the clinical guidelines and clinical practice internationally.

   *Adjustment for COVID-19: The COVID-19 pandemic has resulted in unseasonal RSV and bronchiolitis seasons. As such, adjustments will be made to study recruitment to ensure recruitment occurs during peak RSV times. In order to achieve this aim, the study may in some sites recruit for 12 months of the year.
2. Age 60 days to less than 12 months. Children younger than 60 days will not be enrolled due to the risk of concomitant infection and other issues pertaining to glucocorticoid use in the very young. Children older than 12 months will not be enrolled to minimize the risk of enrolling children with asthma.

Exclusion Criteria:

1. Respiratory distress assessment instrument (RDAI) score of less than or equal to 3. This RDAI will ensure children with very mild respiratory diseases are not enrolled. This is the lower limit of the RDAI range used in CanBEST.
2. Previously known chronic disease that may affect cardiopulmonary status of the patient, such as bronchopulmonary dysplasia currently receiving oxygen, cystic fibrosis, congenital heart disease and immune deficiency. These children may be at higher risk for developing severe illness.
3. Severe respiratory distress evidenced by a sustained pulse rate > 200 beats/min, a sustained respiratory rate > 80 breaths/min, profound lethargy (as deemed by the treating physician), or requiring resuscitation room care. We will exclude these children as they are likely to be admitted due to severity of illness.
4. Presenting with symptoms of apnea prior to enrollment.
5. Treatment with oral, inhaled, or IV corticosteroids within the last 1 week.
6. History of adverse reaction to glucocorticoids.
7. Treatment with any beta-agonists (salbutamol/albuterol or epinephrine/adrenaline) in the ED prior to study enrolment.
8. Presence of varicella or recent (less than 3 weeks) close contact (defined as any household or daycare contact, or greater than 15 minutes of face to face contact, or greater than 1 hour of being in the same dwelling with an individual) without a history of prior infection. These patients are not enrolled to reduce any risk of developing severe varicella with corticosteroid use.
9. Insurmountable language barrier (patient's parent/guardian is unable to understand English or French to give informed consent and participate in follow-up).
10. Any child born at less than 37weeks gestation who is younger than 60 days corrected age. We will not enroll these children to lower any risk of exposing young infants to corticosteroids.
11. Previous enrolment in the trial.
12. Unavailability for follow-up period.
13. Certain admission to hospital.

Ages: 60 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 864 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Admission to hospital for bronchiolitis within 7 days post enrollment | 7 days post enrollment
  1) patient being admitted to inpatient ward, or 2) an ED length of stay 12 hours or greater or 3) a combined ED and observation unit stay of 12 hours or greater.

SECONDARY OUTCOMES:
Admission to hospital for bronchiolitis at the time of the enrollment ED visit | Enrollment visit
  1) patient being admitted to inpatient ward, or 2) an ED length of stay 12 hours or greater or 3) a combined ED and observation unit stay of 12 hours or greater.
All cause admission to Hospital within 21 days following enrollment ED visit | up to 21 days post enrollment
  1) patient being admitted to inpatient ward, or 2) an ED length of stay 12 hours or greater or 3) a combined ED and observation unit stay of 12 hours or greater.
All cause Health care provider visits (including ED visits) by day 21 following enrollment ED | up to 21 days post enrollment
  Visits to ED, other clinic, primary care provider, or any visit to see a nurse or physician following enrollment
Health Care related costs within the 21 days following enrollment ED visits. | up to 21 days post enrollment
  Health care related costs

OTHER OUTCOMES:
Safety outcome 1: Gastrointestinal bleeding | up to 21 days post enrollment
  involving melena or frank blood per rectum (and not attributable to other causes, as determined by the treating physician)
Safety outcome 2: Serious Bacterial Infection | up to 21 days post enrollment
  meningitis, osteomyelitis or septicaemia
Safety outcome 3: Severe Varicella | up to 21 days post enrollment
  All of the following including: arthritis, osteomyelitis, symptomatic hepatitis, pancreatitis, cerebritis, pneumonitis, glomerulonephritis, disseminated intravascular coagulation, thrombo-cytopenia, prolonged vesicular rash (<3 weeks), fasciitis, septicaemia, ocular complications, orchitis, myocarditis, intensive care admission and death
Safety outcome 4: Death | up to 21 days post enrollment
  Death
Exploratory Outcome 1: Admission to hospital for bronchiolitis within 21 days following enrollment ED visit | up to 21 days post enrollment
  1) Patient admitted to inpatient ward, or 2) an ED length of stay 12 hours or greater or 3) a combined ED and observation unit stay of 12 hours or greater.
Exploratory Outcome 2: Admission to ICU within 21 days following enrollment ED visit for bronchiolitis and requiring intubation or continuous positive airway pressure (CPAP) | up to 21 days post enrollment
  Physician admitting patient to ICU for bronchiolitis and requiring oxygen or ventilatory support
Exploratory Outcome 3: All cause admission to hospital with 7 days following enrollment ED visit | up to 7 days post enrollment ED visit
  1) Patient admitted to inpatient ward, or 2) an ED length of stay 12 hours or greater or 3) a combined ED and observation unit stay of 12 hours or greater.
Exploratory Outcome 4: All cause ED visits within 21 days following enrollment ED visit | up to 21 days post enrollment ED
  Visits to the ED after initial enrollment ED visit
Exploratory Outcome 5: Length of stay for the enrollment ED visit (in hours) | Enrollment ED visit
  defined as discharge time minus oral study medication time, for participants discharged at the enrollment ED
Exploratory Outcome 6: Length of hospital admission for those patients admitted at their enrollment visit | Admissions at enrollment ED visit
  time of hospital discharge minus the time of oral study medication
Exploratory Outcome 7: Resolution of symptoms as documented on a standardized questionnaire during the telephone or email at day 7 and 21 days. | up to 21 days post enrollment
  cough, noisy breathing, respiratory distress, sleep and ability to feed
Exploratory Outcome 8: Out of pocket expenses | up to 21 days post enrollment
  transportation, days of missed work, missed leisure activities
Exploratory Outcome 10: Health care utilization (including ambulatory visits, ED visits, hospitalization) for respiratory illness | Up to 18 years of age
  future health care utilization
Exploratory Outcome 11: Development of respiratory illnesses | Up to 18 years of age
  asthma, wheezing and other respiratory illnesses

CONTACTS AND LOCATIONS:
Overall Officials: Amy Plint, MSc, MD, Principal Investigator — Childrens Hospital of Eastern Ontario (CHEO)
Locations (12):
- Australia (3):
  - Women and Children's Hospital, Adelaide
  - Monash Medical Centre, Melbourne
  - Perth Children's Hospital, Perth
- Canada (6):
  - Children's Hospital of Alberta, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Childrens Hospital at London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justines Hospital, Montreal, Quebec
  - Children's Hospital of Winnipeg, Sherbrook, Winnipeg
- New Zealand (3):
  - Starship Children's Hospital, Auckland
  - Kidz First Hospital, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heath A, Rios D, Vogel KI, Rowe T, Wills-Ibarra N, Oakley E, Offringa M, Pechlivanoglou P, Klassen TP, Dalziel SR, Plint AC; KidsCan Pediatric Emergency Research Canada (PERC) Innovative Pediatric Clinical Trials and Pediatric Research in Emergency Department International Collaborative (PREDICT) BIPED Study Team. A randomised controlled trial comparing epinephrine and dexamethasone to placebo in the treatment of infants with bronchiolitis (BIPED study): a statistical analysis plan. Trials. 2025 Nov 12;26(1):496. doi: 10.1186/s13063-025-09125-w. PMID 41225556
- [Derived] Lan J, Plint AC, Dalziel SR, Klassen TP, Offringa M, Heath A; Pediatric Emergency Research Canada (PERC) KIDSCAN/PREDICT BIPED Study Group. Remote, real-time expert elicitation to determine the prior probability distribution for Bayesian sample size determination in international randomised controlled trials: Bronchiolitis in Infants Placebo Versus Epinephrine and Dexamethasone (BIPED) study. Trials. 2022 Apr 11;23(1):279. doi: 10.1186/s13063-022-06240-w. PMID 35410375